CLINICAL TRIAL: NCT01776710
Title: Development and Piloting of a Pragmatic Structured Education Programme That Promotes Walking in Patients With Intermittent Claudication
Brief Title: Structured EDucation for Rehabilitation in Intermittent Claudication
Acronym: SEDRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other); University of York (Other); University of Stirling (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STH17173
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Intermittent claudication; Behavior therapy; Walking; Exercise; Patient education; Randomized controlled trial
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured education (Experimental): The structured education intervention will comprise a 3-hour education workshop delivered by two trained facilitators and a follow-up telephone call 2 weeks later. The aims of the education programme are to enhance patients' understanding of peripheral arterial disease and intermittent claudication, and to support patients in increasing their daily walking activity. Key behaviour change techniques that will be incorporated will include goal setting, action planning, barrier identification/problem solving, prompt review of behavioural goals, prompt self-monitoring of behaviour, and instructions on how to perform the behaviour.
  Interventions: Behavioral: Structured education
- Standard care control (No Intervention): Standard care will consist of general advice to increase walking and an information sheet on peripheral arterial disease, plus a consultation with a Consultant Vascular Surgeon.

INTERVENTIONS:
Behavioral: Structured education — The structured education intervention will comprise a 3-hour education workshop delivered by two trained facilitators and a follow-up telephone call 2 weeks later. The aims of the education programme are to enhance patients' understanding of peripheral arterial disease and intermittent claudication, and to support patients in increasing their daily walking activity. Key behaviour change techniques that will be incorporated will include goal setting, action planning, barrier identification/problem solving, prompt review of behavioural goals, prompt self-monitoring of behaviour, and instructions on how to perform the behaviour.
  Arms: Structured education

SUMMARY:
A primary therapeutic goal for patients with intermittent claudication (IC) is to regain lost physical function through exercise rehabilitation. Supervised exercise programmes can markedly improve walking capacity, but these are resource intensive, National Health Service provision is limited, and patients cite accessing services as a barrier to participation.

Increasing walking activity via a structured education programme might be a pragmatic solution for improving walking capacity, health and wellbeing in patients with IC; however, further research is needed to substantiate this. Hence, the aim of this project is to develop a pragmatic education programme to increase walking in these patients and to collect data on its feasibility to inform the development of a definitive trial investigating clinical and cost effectiveness.

Focus groups will be conducted to inform the development of the education programme. Programme components will be theoretically-underpinned and evidence-based. The development of the programme will be an iterative process involving pilot work, feedback, evaluation, and revision. The programme will then be assessed in a randomised controlled pilot study with 6-week follow-up (n=30). We will assess the feasibility of the intervention and obtain preliminary data of its impact on important outcomes (daily steps/physical activity, walking capacity, quality of life, illness perceptions).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years with intermittent claudication due to peripheral arterial disease
* Stable disease for >3 months
* Able to provide consent
* Able to read and speak English to a level allowing satisfactory completion of written questionnaires and to participate in the education intervention

Exclusion Criteria:

* Previous endovascular/surgical interventions
* Scheduled endovascular/surgical intervention
* Critical limb ischaemia
* Those whose function is uniquely impaired, e.g. wheelchair-bound patients and patients with lower-extremity amputation(s)
* Presence of contraindications to exercise or co-morbidities that limit exercise performance to a greater extent than the intermittent claudication (e.g. severe arthritis)
* Major surgery, myocardial infarction or stroke/transient ischemic attack in the previous 6 months
* Patients who already perform greater than 30 min of structured exercise three times weekly (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 weeks
  The feasibility of the structured education programme will be assessed in terms of recruitment, retention, compliance and acceptability, the latter of which will assessed via participant interviews.

SECONDARY OUTCOMES:
Daily steps and physical activity | 6 weeks
  Daily steps and physical activity will be measured objectively using Actigraph GT3X+ accelerometers. Participants will wear this device for seven consecutive days. A 'valid day' will consist of at least 10 h of accelerometer movement data and participants with less than 4 days (3 weekdays and 1 weekend day) of valid wear will be excluded from the analysis.
Claudication onset and maximum walking distances | 6 weeks
  Claudication onset and maximum walking distances will be assessed using an incremental treadmill test and a 6-min corridor walking test. The treadmill protocol will start at 3.2 km/hr, 0% grade for 2 minutes, with 2% increases in grade every 2 minutes up to 18%, which is maintained until the patient needs to stop.
Self-reported ambulatory ability | 6 weeks
  Self-reported ambulatory ability will be assessed using the Walking Impairment Questionnaire and the Estimation of Ambulatory Capacity by History Questionnaire.
Health-related quality of life | 6 weeks
  Health-related quality of life will be assessed using the EuroQol EQ5D-5L questionnaire, and the Intermittent Claudication Questionnaire
Psychological constructs representing the key mediators of behaviour change | 6 weeks
  Psychological constructs representing the key mediators of behaviour change suggested by the underpinning theories will also be assessed including: Illness perceptions (The Brief Illness Perception Questionnaire), walking self-efficacy, barrier self-efficacy, and action planning.

OTHER OUTCOMES:
Participants' experiences | 6 weeks
  We aim to explore participants' experiences at the end of the 6-week follow-up visit via a one-to-one semi-structured interview (up to 1 hour; audio-recorded and transcribed). Issues discussed will include quality of life, function and attitudes to walking, the acceptability of the intervention and outcomes measures, and the strength of preferences for either the intervention or control arms.

CONTACTS AND LOCATIONS:
Overall Officials: Garry A Tew, PhD, Principal Investigator — University of York
Locations (1):
- Department of Health Sciences, University of York, York, North Yorkshire, United Kingdom